CLINICAL TRIAL: NCT00506857
Title: Phase I/II Trial of Fludarabine in Combination With Intravenous Busulfan and Allogeneic Progenitor Cell Support for Patients With Hematologic Malignancies
Brief Title: Phase I/II Trial of Fludarabine Plus Busulfan and Allogeneic Progenitor Cell Support
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM99-251
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-01

CONDITIONS: Hematologic Malignancies
Keywords: Hematologic Malignancies; Blood And Marrow Transplantation; Leukemia; MDS; Lymphoma; Myeloma; Fludarabine; Fludara; Fludarabine Phosphate; Busulfan; Busulfex; Myleran; Progenitor Cell Transplantation; Granulocyte colony stimulating factor; G-CSF; Apheresis; Blood cell infusion
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasms, Plasma Cell | interventions — Busulfan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busulfan + Fludarabine (Experimental): Busulfan starting 0.8 mg/kg by vein (IV) every 6 hours for 12 doses; Fludarabine 30 mg/m^2 IV daily for 4 days.
  Interventions: Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Busulfan — Starting Dose 0.8 mg/kg by vein every 6 hours x 12 doses.
  Other Names: Busulfex; Myleran
Drug: Fludarabine — 30 mg/m^2 by vein daily x 4 days.
  Other Names: Fludarabine phosphate; Fludara

SUMMARY:
Objectives:

1. To determine the relative toxicities, engraftment potential, kinetics of engraftment, degree of chimerism and disease control achieved with the combination of fludarabine and busulfan at different dose levels and different dose schedules in patients undergoing allogeneic stem cell transplant (SCT).
2. Determine pharmacokinetics, and toxicity of intravenous busulfan given at equal total dose levels given four times daily, or once daily.
3. In vivo determination of fludarabine inhibitory effects on DNA repair.

DETAILED DESCRIPTION:
Treatment: Participants will have blood tests and bone marrow tests as well as tests to check lung, heart, kidney, and liver functions. Participants will receive busulfan by vein for 2 to 4 days depending on their age and medical condition. All participants will receive fludarabine which will be given over 4 days. Participants undergoing unmatched or matched unrelated donors will receive ATG over 4 days to help with the engraftment of the donor progenitor cells. All drugs are given through the vein daily.

The donor blood cells will be taken from the donor through a process known as apheresis. This will occur after the donor has received 2 days of granulocyte colony stimulating factor (G-CSF) to increase her/his white cell count. The G-CSF will also increase the number of very immature (stem cells) that are to be collected. Apheresis is similar to a platelet donation, but white cells and stem cells are collected instead. About 3 to 5 apheresis procedures will be needed to get enough cells for infusion. If apheresis is not used, donor bone marrow will be taken under general anesthesia.

After the participants receives the donor stem cells, the stem cells divide and reconstitute bone marrow function, blood function, and immunity. The donor stem cells are given after the chemotherapy to shorten the period of low blood counts. They are also given at this time to achieve an antileukemic effect whereby the donor immune cells will recognize the participant's leukemia as "foreign" and prevent its recurrence. A small amount of donor cells will be kept for infusion on a future date (usually 3 and 6 months post transplant) to try to prevent the disease from coming back.

During the 4 to 8 weeks following blood cell infusion, participants will need frequent blood tests to monitor their counts and blood chemistries. Participants will need frequent blood transfusion and may have to be admitted to the hospital to receive antibiotics if they develop fever. Bone marrow will be examined frequently beginning four weeks after treatment to check response. Participants that achieve normal bone marrow and blood counts will be evaluated to determine the most appropriate form of future therapy. Participants who fail to respond to treatment will be offered other therapies.

This is an investigational study. All through all drugs are commercially available. Up to 140 participants will take part in this study. All will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Less than physiologic 75 years of age.
2. Interferon resistant late chronic phase CML not eligible for a protocol of higher priority.
3. Accelerated/Blastic Phase CML.
4. Acute leukemia or Intermediate to High Risk MDS according to the IPPS.
5. Any Lymphoma or Myeloma beyond CR1 ineligible for a protocol of higher priority.
6. Patients must have an HLA compatible donor willing to donate either peripheral blood or bone marrow progenitor cells.
7. Both patients and donor must sign written informed consents.

Exclusion Criteria:

1. Uncontrolled infection
2. Bilirubin >3.0
3. Creatinine >2.5
4. Performance Status >Zubrod 2

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2003 to August 2011. All recruitment was done at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 82 participants enrolled, two (2) participants were excluded from the trial before starting treatment.
Period: Overall Study
Arm/Group | Busulfan + Fludarabine
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan + Fludarabine
Number analyzed (Participants) | 80
Age Continuous [Median (Full Range); unit: years] | 56 [10 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 54
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Continual reassessment method (four times a day) used to determine an MTD, with a target toxicity probability of 20%, where "toxicity" is defined as grade 3 or 4 conventional toxicity [National Cancer Institute Common Toxicity Criteria (NCI-CTC)]. Participant evaluation in a cohort with each modality is 30 days.
Time Frame: 1 month
Population: Analysis was per protocol.
Measure: Number; unit: mg/kg
Arm/Group | Busulfan + Fludarabine
Number analyzed (Participants) | 80
mg/kg | 11.2

2. Secondary Outcome: Number of Participants With Graft Versus Host Disease (GVHD)
Description: Tacrolimus and Methotrexate used for acute graft versus host disease (aGVHD) prophylaxis, clinical grading AGVHD criteria (Days 1-100): Grade 1: + to ++ skin rash; no gut involvement; no decrease in clinical performance status; Grade 2: + to +++ skin rash; + gut involvement and/or + liver involvement; mild decrease in performance status; Grade 3: ++ to +++ skin rash; ++ to +++ gut involvement and/or ++ to ++++ liver involvement; marked decrease in performance status; Grade 4: Similar to Grade 3 with ++ to ++++ organ involvement and extreme decrease in performance status.
Time Frame: 5 years
Population: Analysis was per protocol for 73 patients out of 80 patients due to 3 early deaths and 4 non engraftments.
Measure: Number; unit: Participants
Groups:
- Tacrolimus + Methotrexate: Busulfan starting 0.8 mg/kg by vein (IV) every 6 hours for 12 doses; Fludarabine 30 mg/m^2 IV daily for 4 days.
Arm/Group | Tacrolimus + Methotrexate
Number analyzed (Participants) | 73
Participants
  Grade 2 | 18
  Grade 3-4 | 8

ADVERSE EVENTS:
Time Frame: March 2000 to December 2004 (4 years, 8 months)
Arm/Group | Busulfan + Fludarabine
Serious Adverse Events (participants affected / at risk) | 72/80
Other Adverse Events (participants affected / at risk) | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Busulfan + Fludarabine (N=80)
Graft failure (Blood and lymphatic system disorders) | 2
Infections (Infections and infestations) | 12
Diffuse alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7
Death (General disorders) | 8
Chronic Graft versus Host Disease (General disorders) | 8/73
Mucositis (Gastrointestinal disorders) | 1
Epistaxis (Gastrointestinal disorders) | 3
Acute Graft versus Host Disease (General disorders) | 26/73
Elevated alanine aminotransferase (Hepatobiliary disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan + Fludarabine (N=80)
Diarrhea (Gastrointestinal disorders) | 30
Nausea (Gastrointestinal disorders) | 39
Elevated Creatinine (Renal and urinary disorders) | 32
Hemorrhagic cystitis (Renal and urinary disorders) | 2
Elevated alkaline phosphate (Hepatobiliary disorders) | 3
Altered mental status (Nervous system disorders) | 2
Occular (Eye disorders) | 5
Fever (General disorders) | 5
Lethargy (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 6
Stomatitis/Esophagitis (Gastrointestinal disorders) | 23
Hepatotoxicity (Hepatobiliary disorders) | 15
Elevated alanine aminotransferase (Hepatobiliary disorders) | 27 — Diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No